CLINICAL TRIAL: NCT05999058
Title: Clinical Characteristics and Treatment Outcomes of Nasolacrimal Duct Obstruction Using Dacryoendoscopy
Brief Title: Clinical Study of Lacrimal Drainage Obstruction Diseases Using Dacryoendoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY-2023038
Record Dates: First submitted 2023-08-13; First posted 2023-08-21 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Lacrimal Duct Obstruction
Keywords: Lacrimal Duct Obstruction; Dacryoendoscopy; Dacryoplasty
MeSH Terms: conditions — Lacrimal Duct Obstruction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Active Comparator): group A higher nasolacrimal duct obstruction
  Interventions: Procedure: Dacryoendoscopic-assisted laser dacryoplasty with silicone intubation
- group B (Experimental): group B: lower nasolacrimal duct obstruction
  Interventions: Procedure: Dacryoendoscopic-assisted laser dacryoplasty with silicone intubation
- group C (Experimental): group C: nasolacrimal duct stenosis
  Interventions: Procedure: Dacryoendoscopic-assisted laser dacryoplasty with silicone intubation

INTERVENTIONS:
Procedure: Dacryoendoscopic-assisted laser dacryoplasty with silicone intubation — The dacryoendoscopy was inserted into the lacrimal duct through the upper or lower lacrimal punctum. When the dacryoendoscopy reached the postsaccal obstruction, laser dacryoplasty (FOX diode laser, A.R.C. Laser, Nürnberg, Germany) was performed by widening the stenotic or obstructed section. After removing the dacryoendoscopy, a silicone tube inserted into lacrimal passage. Double bicanalicular silicone intubation was performed as previously described.

SUMMARY:
Nasolacrimal duct obstruction (NLDO) can manifest as epiphora or recurrent infections with mucopurulent discharge and may even cause social embarrassment. Dacryoendoscopic-assisted laser dacryoplasty with silicone intubation (DLDI) offers direct therapy to the obstructed site, leading to minimal collateral damage external to the target zone. Although the silicone intubation using dacryoendoscopy has increased the success rates, the success rates vary from a low of 51% to a high of 90%. The difference in success rates seems to depend on the site of obstruction, differences in the surgical technique, stringency of definitions of success, and duration of follow-up. The aim of our study was to report the results of DLDI for the management of NLDO, and to identify factors associated with DLDI failure.

DETAILED DESCRIPTION:
Lacrimal drainage obstruction can manifest as epiphora or recurrent infections with mucopurulent discharge and may even cause social embarrassment. Obstruction can occur at any level along the lacrimal drainage system: punctum, canaliculus, nasolacrimal duct, or nasal ostium. It is seen more often in females, especially in postmenopausal women. The etiopathogenesis of lacrimal passage obstruction appears to be multifactorial. Chronic inflammation has been suggested to be the most causal. Dacryocystorhinostomy (DCR) is a standard surgical procedure used to treat nasolacrimal duct obstruction (NLDO), with a reported success rate of more than 90%.

Knowledge concerning the morphological characteristics of lacrimal passage obstruction using traditional diagnostic methods (e.g., lacrimal irrigation, probing, dacryocystography) is limited. Dacryoendoscopy was originally described in 1979 and has recently matured for use in lacrimal drainage system imaging. It has been proved to be a useful instrument not only for understanding differences in the etiology of obstructions but also for treating LD obstructions. On the other hand, semiconductor diode laser can achieve more effective tissue dissection than direct probing technique with minimal hemorrhage and improved intraoperative view. Hence, dacryoendoscopic-assisted laser dacryoplasty with silicone intubation (DLDI) offers direct therapy to the obstructed site, leading to minimal collateral damage external to the target zone. In addition, this procedure can be performed under local anesthesia as an outpatient procedure in the office, and it has advantages such as short surgery time and less risk of bleeding during surgery, resulting in its increasingly widespread use in China. Although the silicone intubation using dacryoendoscopy has increased the success rates, the success rates vary from a low of 51% to a high of 90%. The difference in success rates seems to depend on the site of obstruction, differences in the surgical technique, stringency of definitions of success, and duration of follow-up.

A greater understanding of factors associated with treatment failure may allow us to glean insights regarding patient selection and ultimately improve treatment outcome. The aim of our study was to report the results of DLDI for the management of NLDO, and to identify factors associated with DLDI failure.

ELIGIBILITY:
Inclusion Criteria:

(1) confirmed diagnosis of nasolacrimal duct obstruction or stenosis, based on dacryoendoscopic examination with or without radiologic confirmation on dacryocystogram; (2) recurrent or persistent and symptomatic epiphora; (3) follow-up of longer than 6 months after removal of the silicone stent.

Exclusion Criteria:

(1) congenital or traumatic lacrimal duct obstruction; (2) previous acute dacryocystitis; (3) facial nerve palsy; (4) lower eyelid or punctal malposition or laxity of sufficient severity to contribute to epiphora; (5) previous dacryocystorhinostomy; (6) incomplete medical records.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 522 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Cumulative success rate | 2 years
  The main outcome measure was the cumulative success rate of DLDI within 2 years follow-up of obtained using the Kaplan-Meier estimator.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li H, Li J, Zhang L, Yang L, Zhao Y, Zhao H, Pan Y. Clinical outcomes and prognostic factors in patients with nasolacrimal duct obstruction or stenosis using dacryoendoscopy. BMJ Open Ophthalmol. 2024 Oct 31;9(1):e001743. doi: 10.1136/bmjophth-2024-001743. PMID 39486803